CLINICAL TRIAL: NCT03651531
Title: Comparison of Insulin Alone to Insulin With Metformin to Treat Gestational Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial halted early due to limited ability to recruit participants
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1099865-3
Record Dates: First submitted 2018-06-12; First posted 2018-08-29 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Gestational Diabetes
Keywords: metformin
MeSH Terms: conditions — Diabetes, Gestational | interventions — Insulin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- insulin (Active Comparator)
  Interventions: Drug: Insulin
- insulin and metformin (Active Comparator)
  Interventions: Drug: Insulin; Drug: Metformin

INTERVENTIONS:
Drug: Insulin — Weight based insulin will be calculated using 0.7 units/kg/day in the first trimester, 0.8 units/kg/day in the second trimester and 1 units/kg/day in the third trimester. This total insulin will then be divided into short acting insulin and intermediate acting insulin per provider discretion.
Drug: Metformin — Will be initiated at dose of 500 mg twice daily. If glycemic control is suboptimal, the dose of metformin will be increased to 1000 mg twice a day. Metformin will be titrated prior to increases in insulin.
  Arms: insulin and metformin

SUMMARY:
This study is a prospective, unmasked randomized clinical trial comparing the use of insulin vs combination insulin and metformin for treatment in women diagnosed with gestational diabetes mellitus (GDM). The investigator's hypothesis is that the combination of metformin and insulin will be superior to insulin alone to achieve tight glucose control during pregnancy.

DETAILED DESCRIPTION:
The objective of this study is to compare the effectiveness of insulin alone vs the combination of insulin and metformin in treating patients with gestational diabetes (GDM). Currently, outside of pregnancy, the treatment of type 2 diabetes mellitus (T2DM) with both metformin and insulin is superior to using insulin alone. In pregnancy, insulin alone has traditionally been used, though some advocate the use of metformin alone as primary therapy. There have been no trials published to date specifically comparing combination therapy to insulin alone. Our hypothesis is that the combination of metformin and insulin will improve overall control of blood glucose, the improvement of which has been demonstrated to improve maternal and neonatal outcomes. Control of blood glucose will be determined by hemoglobin A1c at the time of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write English and/or Spanish and give written consent
* Diagnosis of GDM, defined as an abnormal glucose tolerance test performed after 12 weeks gestation using 1 of the 2 criteria below:
* 50 gram 1 hour oral diabetes screening testing yielding a result of > 200 mg/dL
* A 100 gram 3 hour oral glucose tolerance testing yielding >2 abnormal values (normal values defined as fasting blood glucose < 95, 1 hour < 180, 2 hour < 155 and 3 hour < 140)
* Singleton gestation
* Gestational age between 12 and 34 weeks and 6 days determined by last menstrual period (LMP) confirmed by ultrasound using criteria set forth by the ACOG (Committee on Obstetric Practice). If LMP is unknown then gestational age must be set by ultrasound prior to 20 weeks gestation.

Exclusion Criteria:

* Pre-existing DM either by diagnosis preceding pregnancy or hemoglobin A1c >6.5 collected during the current pregnancy
* Uncontrolled chronic hypertension, as this may alter maternal and perinatal outcomes measured.
* Multiple gestations
* Major fetal anomalies anticipated to require NICU admission
* Contraindication to metformin (allergy, history of lactic acidosis, pre-existing renal disease (Cr >1.5 mg/dL), active liver disease, current alcohol abuse).
* Vitamin B12 deficiency, as metformin reduces intestinal absorption of vitamin B12
* Medications known to effect glucose metabolism other than insulin and metformin as this may mask any effect between the two treatments.
* Known inability to tolerate metformin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Hgb A1c | collected at the time of delivery
  Hgb A1c test

SECONDARY OUTCOMES:
Total daily dose of insulin | Will be recorded on hospital admission for delivery
  Total daily dose of insulin at the end of pregnancy
Glucose control | patients will collect glucose values fasting and 2 hrs postprandial every day from enrollment until delivery.
  Average of fasting and 2 hour postprandial glucose values
Incidence of maternal hypoglycemia | patients will be screened weekly for episodes of hypoglycemia until delivery
  episodes of maternal hypoglycemia defined as glucose ≤70 mg/dL
Change in hemoglobin A1c over the course of the pregnancy | hemoglobin A1c will be collected at delivery (per above) and comparison performed after collection
  If baseline hemoglobin A1c was collected as part of routine care prior to enrollment, this value will be compared to the hemoglobin A1c collected at delivery
Incidence of maternal side effects | Will be assessed weekly until delivery
  maternal reported medication side effects (i.e. nausea, vomiting, diarrhea)
Treatment acceptability | Will be collected postpartum after delivery
  determined using Diabetes Treatment Satisfaction Questionnaire. Survey includes 8 questions that are answered on a scale of 0-6; 0 indicating the least and 6 the highest level of satisfaction. The individual questions will be compared. Total satisfaction will also be compared by summing the responses to all 8 questions on a composite scale of 0-48
Maternal weight gain | This will be calculated as the difference from the weight measured at the inital prenatal visit (the specific timing of which is patient dependant) and at the time of admission for delivery
  weight gain through pregnancy
Incidence of hypertensive disorder of pregnancy | from enrollment through study completion (30 days after delivery)
  gestational HTN, superimposed pre-eclampsia, pre-eclampsia-eclampsia
Incidence of composite of adverse maternal outcomes | from enrollment through study completion (30 days after delivery)
  death, ICU admission, postpartum hemorrhage, blood transfusion, organ failure, chorioamnionitis/endometritis
Breast feeding status | Will be recorded at the time of hospital discharge after delivery (typically 2-4 days after delivery)
  Whether patient is breast feeding or bottle feeding upon discharge from the hospital after delivery
Mode of delivery | recorded at time of delivery
  Mode of delivery
Gestational age at delivery | recorded at time of delivery
  Gestational age at delivery
Infant birthweight (using age/sex matched percentiles) | measured at time of birth
  Infant birthweight (using age/sex matched percentiles)
Incidence of composite neonatal morbidity | from delivery through study completion (30 days after delivery)
  Presence of any of the following: NICU admission, hypoglycemia, hyperbilirubinemia, birth trauma, stillbirth, respiratory distress syndrome, sepsis, neonatal death prior to discharge, 5 minute Apgar score < 7, umbilical artery cord pH <7.10
Incidence neonatal hypoglycemia | from delivery through study completion (30 days after delivery)
  hypoglycemia requiring intravenous treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nau, MD, Principal Investigator — Women & Infants Hospital; Erika Werner, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee Opinion No 700: Methods for Estimating the Due Date. Obstet Gynecol. 2017 May;129(5):e150-e154. doi: 10.1097/AOG.0000000000002046. PMID 28426621